CLINICAL TRIAL: NCT01039571
Title: Prospective Randomized Case-controlled Blinded Study of Single Versus Double Row Suture Anchor Repair in Medium to Large Rotator Cuff Tears
Brief Title: Single Versus Double Row Suture Anchor Repair in Medium to Large Rotator Cuff Tears
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Samsung Medical Center, Samsung Medical Center
Other Study IDs: 2005-12-005
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff tear; arthroscopic repair; single row repair; double row repair; retear rate
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: double row repair — double row repair for torn rotator cuff were performed to compare with the conventional single row repair
  Other Names: dual row repair

SUMMARY:
The purpose of this study is to determine whether double row repair is better in healing than traditional single row repair in arthroscopic rotator cuff repair.

Our null hypothesis is there are no differences in clinical and structural results

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff tears
* tear size between 2cm~4cm

Exclusion Criteria:

* Subscapularis tear requiring repair
* open repair
* any prior history of surgery on the affected shoulder
* any fracture history around shoulder girdle(clavicle, humerus, acromion)
* glenohumeral joint arthritis
* inflammatory arthropathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rotator cuff tear patients
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2005-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Retear rate in each group(single row repair group and double row repair group) | MRI after 6 months from surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Grasso A, Milano G, Salvatore M, Falcone G, Deriu L, Fabbriciani C. Single-row versus double-row arthroscopic rotator cuff repair: a prospective randomized clinical study. Arthroscopy. 2009 Jan;25(1):4-12. doi: 10.1016/j.arthro.2008.09.018. Epub 2008 Nov 1. PMID 19111212
- [Background] Burks RT, Crim J, Brown N, Fink B, Greis PE. A prospective randomized clinical trial comparing arthroscopic single- and double-row rotator cuff repair: magnetic resonance imaging and early clinical evaluation. Am J Sports Med. 2009 Apr;37(4):674-82. doi: 10.1177/0363546508328115. Epub 2009 Feb 9. PMID 19204365
- [Background] Franceschi F, Ruzzini L, Longo UG, Martina FM, Zobel BB, Maffulli N, Denaro V. Equivalent clinical results of arthroscopic single-row and double-row suture anchor repair for rotator cuff tears: a randomized controlled trial. Am J Sports Med. 2007 Aug;35(8):1254-60. doi: 10.1177/0363546507302218. Epub 2007 Jun 6. PMID 17554104
- [Background] Charousset C, Grimberg J, Duranthon LD, Bellaiche L, Petrover D. Can a double-row anchorage technique improve tendon healing in arthroscopic rotator cuff repair?: A prospective, nonrandomized, comparative study of double-row and single-row anchorage techniques with computed tomographic arthrography tendon healing assessment. Am J Sports Med. 2007 Aug;35(8):1247-53. doi: 10.1177/0363546507301661. Epub 2007 Apr 23. PMID 17452513
- [Background] Mazzocca AD, Millett PJ, Guanche CA, Santangelo SA, Arciero RA. Arthroscopic single-row versus double-row suture anchor rotator cuff repair. Am J Sports Med. 2005 Dec;33(12):1861-8. doi: 10.1177/0363546505279575. Epub 2005 Oct 6. PMID 16210578
- [Background] Park JY, Lhee SH, Choi JH, Park HK, Yu JW, Seo JB. Comparison of the clinical outcomes of single- and double-row repairs in rotator cuff tears. Am J Sports Med. 2008 Jul;36(7):1310-6. doi: 10.1177/0363546508315039. Epub 2008 Apr 15. PMID 18413680